CLINICAL TRIAL: NCT06046053
Title: MATRIX-002: Trial to Assess Acceptability and Safety of Two Placebo Prototype Vaginal Films
Brief Title: MATRIX-002: Trial to Assess Acceptability and Safety of Two Placebo Vaginal Films
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rohan, Lisa, PhD (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Katherine Bunge, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY23040051
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Safety; Acceptability; Usability
Keywords: Vagina; Film; Placebo

STUDY DESIGN:
Intervention Model Description: Participants will be randomized (1:1) to insert either placebo vaginal film A or placebo vaginal film B once monthly for two months. Films A and B are 2" x 2" in size and differ only by shape (square versus rounded corners).
Masking Description: Since the two films will differ by shape, masking is not possible once the product is removed from packaging for the participant and clinicians assessing the clinical outcomes. However, the assessors of the vaginal microenvironment endpoints will be masked as to product assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo Vaginal Film with Square Corners (Experimental): A single 2" x 2" placebo vaginal film with square corners, inserted intravaginally once monthly for two months.
  Interventions: Drug: Placebo Vaginal Film with Square Corners
- Placebo Vaginal Film with Rounded Corners (Experimental): A single 2" x 2" placebo vaginal film with rounded corners, inserted intravaginally once monthly for two months
  Interventions: Drug: Placebo Vaginal Film with Rounded Corners

INTERVENTIONS:
Drug: Placebo Vaginal Film with Square Corners — 2" x 2" placebo vaginal film with square corners
  Arms: Placebo Vaginal Film with Square Corners
Drug: Placebo Vaginal Film with Rounded Corners — 2" x 2" placebo vaginal film with rounded corners
  Arms: Placebo Vaginal Film with Rounded Corners

SUMMARY:
This study will enroll approximately 100 HIV-negative persons, aged18-45 years, and assigned female sex at birth from sites in the United States, Kenya, South Africa, and Zimbabwe. The study will assess the acceptability and safety of two placebo vaginal films. The placebo films do not contain any active medication, are the same size, but differ by shape (square versus rounded corners). Participants will be randomly assigned to one of the two films and asked to use (self-insert) the assigned film two times (approximately one month apart). Participants will be asked to refrain from sexual activity during the first month of use and may resume usual sexual activity during the second month of use. The study involves answering questions, undergoing pelvic examinations, and collecting blood and vaginal fluid samples. The study involves a total of 10 visits/contacts, including in person visits and telephone calls over approximately 9 weeks. In addition, both participants and approximately 30 of their sexual partners will be asked to take part in in depth interviews to further assess acceptability, attitudes, and experiences with film use to gauge interest in the future use of vaginal films as a HIV prevention option.

DETAILED DESCRIPTION:
The goal of this randomized, clinical trial is to compare two placebo vaginal films in HIV seronegative adult (18-45 years old) persons assigned female sex at birth who are at low risk of acquiring HIV infection, and sexual partners of evaluable participants. Participants will be recruited from five sites, one in the US and four is sub-Saharan Africa. Approximately 100 participants will be randomized (1:1), stratified by site, to insert either placebo vaginal film A or placebo vaginal film B, which differ only by shape, once monthly for two months. Participants will be asked to refrain from sexual activity during the first month of use and may resume usual sexual activity during the second month of use after insertion of the second film which will be the same film they were assigned to use during the first month. Differences in safety, acceptability, usability, social harms and benefits, and vaginal microenvironment between the two films and the two study phases (i.e., with and without sexual abstinence requirement) will be assessed. In addition, both participants and approximately 30 sexual partners of evaluable participants will be asked to take part in in depth interviews to further assess acceptability, attitudes, and experiences with film use to gauge interest in the future use of vaginal films as a HIV prevention option.

ELIGIBILITY:
Inclusion Criteria:

* Assigned female sex at birth.
* Able and willing to provide written informed consent to be screened for and enrolled in MATRIX-002 in one of the study languages.
* Able and willing to provide adequate contact/locator information.
* Able and willing to comply with all protocol requirements, including:

  * Abstaining from all receptive sexual intercourse (vaginal, anal, digital, oral) for the first month of product use.
  * Abstaining from using other intravaginal products for the first month of product use.
  * Abstaining from engaging in intravaginal practices for the first month of product use.
  * Refraining from participation in other research studies for the duration of the study unless approved by the Protocol Safety Review Team.
  * Responding to scheduled phone/short message service contacts.
  * Attending all clinic follow-up visits.
* HIV-uninfected based on testing performed at Screening and Enrollment.
* Per participant report, if in a relationship, must be in a mutually monogamous relationship with a partner who is not known to be HIV positive or to currently have a sexually transmitted infection.
* Negative urine pregnancy test at Screening and Enrollment.
* Participants over the age of 21 (inclusive) must have documentation of a Grade 0 Pap smear within the past 3 years prior to Enrollment, or a Grade 1 Pap smear at Screening with no treatment required, per the Female Genital Grading Table for Use in Microbicide Studies Addendum 1 (Dated November 2007) to the DAIDS Table for Grading Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017.
* Protected from pregnancy starting two weeks before Screening and continuing for the duration of study participation by an effective contraceptive method; effective methods include:

  * Hormonal methods except vaginal rings
  * Copper intrauterine device
  * Sterilization of participant
  * Correct and consistent condom use (for US site only)
  * Abstinence from penile-vaginal intercourse

Inclusion Criteria for Sexual Partners:

* Identifies as a sexual partner of a MATRIX-002 participant.
* Identified by participant as a sexual partner during MATRIX-002 for whom the participant has given permission to contact.
* Able and willing to provide written informed consent in one of the study languages.
* Able and willing to complete the required study procedures.
* Must be 18 years old or above at the time of their study participation.

Exclusion Criteria:

* Per participant report at Screening and Enrollment, intends to do any of the following during the study participation period:

  * Become pregnant.
  * Breastfeed.
  * Relocate away from the study site.
  * Travel away from the study site for a time period that would interfere with product resupply and/or study participation.
* Positive HIV test at Screening or Enrollment.
* Positive test for Trichomonas vaginalis, Neisseria gonorrhea, Chlamydia trachomatis, or Treponema pallidum (Syphilis) at Screening or (per participant report) treated for potential sexually transmitted infection within past 12 months.
* Diagnosed with urinary tract infection, pelvic inflammatory disease, or reproductive tract infection requiring treatment per WHO guidelines at Enrollment.
* Clinically apparent Grade 2 or higher pelvic exam finding per the DAIDS Table for Grading Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 and/or Addenda 1 (Female Genital Grading Table for Use in Microbicide Studies [Dated November 2007]) at Enrollment.
* Participant report and/or clinical evidence of any of the following:

  * Known adverse reaction to any of the study product materials (ever).
  * Hysterectomy.
  * Surgical procedure involving the pelvis in the 30 days prior to Enrollment.
  * Use of diaphragm, NuvaRing, or (for African sites only) spermicide for contraception in the two weeks prior to Screening.
  * Antibiotic or antifungal (oral or intravaginal) therapy within 7 days of Enrollment.
  * Prior use of post-exposure prophylaxis or oral pre-exposure prophylaxis (including emtricitabine/disoproxil fumarate) in the 4 weeks prior to Screening or any prior use of long-acting systemic pre-exposure prophylaxis (including cabotegravir or islatravir).
  * Use of any of the following in the 12 months prior to Screening: stimulants (cocaine [including crack], methamphetamine, or non-physician prescribed pharmaceutical-grade stimulants), or inhaled nitrates, or illicit injection drug use of any kind.
  * At Screening or Enrollment, as determined by the Investigator of Record/designee, has any significant uncontrolled active or chronic cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, respiratory, immunologic disorder or infectious disease.
* Has any of the following laboratory abnormalities at Screening:

  * Grade 2 or higher Aspartate aminotransferase, alanine transaminase, creatinine, or Hemoglobin per the DAIDS Table for Grading Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017.
* Has any other condition that, in the opinion of the Investigator of record/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2023-10-18 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Mean Satisfaction with Placebo Vaginal Film Use | Through study completion, approximately 9 weeks
  Satisfaction will be assessed using a 10-point Likert scale with 0 being the least satisfied and 10 being the most satisfied

SECONDARY OUTCOMES:
Number of Participants with Genitourinary Grade 2 or Higher Adverse Events | Through study completion, approximately 9 weeks
  Number of participants with genitourinary Grade 2 or higher Adverse Events deemed related to placebo vaginal film use
Number of Participants that Correctly Inserted Vaginal Film | Through study completion, approximately 9 weeks
  Number of participants with clinically assessed proper insertion (more than half of the vaginal film proximal to introitus).

OTHER OUTCOMES:
Mean Change in Vaginal pH | Through study completion, approximately 9 weeks
  Mean change from baseline in vaginal pH and after 1-month of film use during the two study phases (i.e., with and without sexual abstinence requirement).
Mean Change in Nugent Score | Through study completion, approximately 9 weeks
  Mean change in the Nugent score as determined from vaginal smears. Nugent scores range from 0 to 10; 0 indicates a Lactobacillus-dominant microbiome while a score of 10 indicates a microbiome dominated by bacterial vaginosis-associated bacteria. Mean change will be assessed from baseline and after 1-month of film use during the two study phases (i.e., with and without sexual abstinence requirement).

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Bunge, MD, Principal Investigator — University of Pittsburgh
Locations (5):
- Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States
- Kenya Medical Research Institute, Nairobi, Kenya
- South Africa (2):
  - Wits Reproductive Health and HIV Institute, Hillbrow, Johannesburg
  - The Aurum Institute, Klerksdorp, North West
- Harare Health and Research Consortium, Chitungwiza, Zimbabwe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Acceptability Study of Vaginal Films for HIV Prevention (FACE). https://clinicaltrials.gov/ct2/show/NCT01231763?term=NCT01231763&draw=2&rank=1. Accessed February 23, 2023.
- [Background] Musara P, Milford C, Shapley-Quinn MK, Weinrib R, Mutero P, Odoom E, Mgodi NM, Chirenje ZM, Hanif H, Clark MR, Smit J, van der Straten A, Montgomery ET; Quatro Study Team. Preferences and Acceptability of Vaginal Delivery Forms for HIV Prevention Among Women, Male Partners and Key Informants in South Africa and Zimbabwe: Qualitative Findings. AIDS Behav. 2021 Jan;25(1):124-138. doi: 10.1007/s10461-020-02949-4. PMID 32588257
- [Background] Guthrie KM, Rohan L, Rosen RK, Vargas SE, Shaw JG, Katz D, Kojic EM, Ham AS, Friend D, Buckheit KW, Buckheit RW Jr. Vaginal film for prevention of HIV: using visual and tactile evaluations among potential users to inform product design. Pharm Dev Technol. 2018 Mar;23(3):311-314. doi: 10.1080/10837450.2017.1339085. Epub 2017 Jun 21. PMID 28592183

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-24): https://cdn.clinicaltrials.gov/large-docs/53/NCT06046053/Prot_SAP_000.pdf
  • Informed Consent Form (2024-08-08): https://cdn.clinicaltrials.gov/large-docs/53/NCT06046053/ICF_001.pdf